CLINICAL TRIAL: NCT05270460
Title: A Phase 2A, Placebo-controlled, Randomized, Dose Response Study of the Safety, Pharmacokinetics and Efficacy of PCS12852 on Gastric Emptying Rate Assessed by 13C Spirulina GEBT in Patients With Moderate to Severe Gastroparesis
Brief Title: Safety, PK and Efficacy of PCS12852 on Gastric Emptying Rate in Patients With Moderate to Severe Gastroparesis
Acronym: MOMENTUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCS12852-GP-01
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Gastroparesis
Keywords: Idiopathic Gastroparesis; Diabetic Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PCS12852 0.1mg (Experimental): PCS12852 0.1mg tablet
  Interventions: Drug: PCS12852
- PCS12852 0.5mg (Experimental): PCS12852 0.5mg tablet
  Interventions: Drug: PCS12852
- Placebo (Placebo Comparator): Similar in appearance to active study drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PCS12852 — PCS12852 oral tablet administered once daily
  Arms: PCS12852 0.1mg; PCS12852 0.5mg
Drug: Placebo — Placebo comparator oral tablet administered once daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study that will compare the effect of 2 different dosage regimens of PCS12852 on gastric emptying time to placebo in both idiopathic gastroparesis (IG) and diabetic gastroparesis (DG) patients.

ELIGIBILITY:
Inclusion Criteria:

* Has documented diagnosis of moderate to severe DG or IG according to the ANMS GCSI-DD score during the Screening period (score of >2 on average of the screening days).
* Moderate to severe delay in gastric emptying rate as measured by the GEBT at Screening defined as GE half-time (t1/2) ≥ the 80th percentile of normative data as determined by Cairn Diagnostics.
* Male or female patients 18 to 80 years of age, inclusive, at baseline.
* Has continuous moderate to severe symptoms for gastroparesis (that is, chronic postprandial fullness, abdominal pain, postprandial nausea, vomiting, loss of appetite and/or early satiety) as assessed by the investigator for at least the past 3 months.
* Has hemoglobin A1c (BbA1c) < 11%.
* Has Body Mass Index range between 18-40.
* Women of childbearing potential must use one of the following acceptable methods of contraception throughout the study (1 month prior to Screening through 1 month after last dose of study medication): oral contraceptive medication, IUD, hormonal implants, injectable contraceptive methods, double-barrier methods, or tubal ligation.
* Male patients must be willing to use acceptable contraceptive measures such as vasectomy or double-barrier method and refrain from sexual activity with any female who is pregnant or lactating. Female partners of study participants are asked to use acceptable methods of contraception.

Exclusion Criteria:

* Has acute, severe gastroenteritis and pronounced dehydration in the past 48 hours prior to Screening, chronic parenteral feeding or persistent severe vomiting.
* Has known hypersensitivity to Spirulina, egg, milk products or wheat allergens.
* Has a known disturbance of small intestinal absorption, exocrine pancreatic function, liver metabolism or pulmonary function.
* Has a history of anorexia nervosa or bulimia.
* Previous history of bezoars (the presence of retained liquid, bile, or small amounts of poorly organized food residue is permitted).
* Prior surgery involving any gastrointestinal surgery, including the luminal gastrointestinal (GI) tract (cholecystectomy and appendectomy are permitted if performed >3 months prior to baseline GEBT).
* Any abdominal or pelvic surgery within the past 3 months.
* Known history of the following GI conditions: inflammatory bowel disease; irritable bowel syndrome with diarrhea; or any other active disorder that could explain symptoms in the opinion of the investigator.
* Has active diverticulitis, diverticular stricture, and other intestinal strictures.
* Currently taking Glucagon-like peptide-1 (GLP-1) agonists, e.g. exenatide, liraglutide, semaglutide or dulaglutide, or pramlintide.
* Has severe psychiatric illness (including suicidal tendencies or ideation) or neurological illness.
* Use of narcotics/opioids, drugs used to treat gastroparesis within 3 days of the Screening GEBT test.
* Clinically significant cardiac disease including but not limited to unstable angina, acute myocardial infarction within 6 months of baseline, and arrhythmia requiring therapy.
* Patient has QTc interval ≥ 480 milliseconds on Screening ECG.
* History of cerebral hemorrhage, cerebrovascular accident, transient ischemic attack, gastrointestinal bleeding, or retinal hemorrhage within 6 months of baseline.
* Patient has active or history of neoplastic disease (except for adequately treated non-invasive basal cell and/or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) within the past 5 years prior to baseline.
* Presence of clinically significant medical condition(s) including but not limited to: renal, hepatic, cardiovascular, hematological, gastrointestinal, endocrine, pulmonary, neurological, psychiatric, substance abuse, and or any other clinically significant disease or disorder, which in the opinion of the investigator, may put the patient at risk due to participation in the study, influence the results of the study, and/or affect the patient's ability to complete the study.
* History of or current diagnosis of active tuberculosis (TB); undergoing treatment for latent TB infection (LTBI); untreated LTBI (as determined by documented results within 3 months of the Screening Visit of a positive TB skin test with purified protein derivative with induration ≥ 5 mm, a positive QuantiFERON TB test or positive or borderline T-SPOT [Elispot] test); or positive TB test at Screening. Patients with documented completion of appropriate LTBI treatment would not be excluded and are not required to be tested.
* Currently taking known P-gp and BCRP inhibitors or inducers and gastric acid reducing agents. E.g., proton pump inhibitors or H2 receptor antagonists.

Other inclusion/exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - TriWest Research Associates, San Diego, California
  - APF Research, LLC, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - University of Louisville, Louisville, Kentucky
  - Delta Research Partners, Bastrop, Louisiana
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - M3 Wake Research, Raleigh, North Carolina
  - Texas Tech University, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
Started | 9 | 8 | 8
Completed | 9 | 6 | 8
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Early Termination | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 6 | 20
  >=65 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 7 | 22
  Male | 2 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 6 | 14
  Not Hispanic or Latino | 4 | 5 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 7 | 3 | 6 | 16
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 8 | 25
Woman of Childbearing Potential [Count of Participants; unit: Participants] | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Gastric Emptying Rate From Baseline as Determined by the Area Under the Curve (AUC) of the Gastric Emptying Rate
Description: Change from baseline in gastric emptying rate was determined by the AUC by Gastric Emptying Breath Test (GEBT) at Day 28 after administration of PCS12852 or placebo.
Time Frame: ~28 days
Population: The change from baseline to Day 28 in AUC was analyzed using an analysis of covariance (ANCOVA) model with fixed effects for treatment group and gastroparesis type (idiopathic gastroparesis [IG] or diabetic gastroparesis [DG]) and the baseline value as a continuous covariate. Only patients with a baseline and Day 28 value were included in the analysis. The parameters listed are the best comparison of the breath test as opposed to individual timepoints.
Measure: Least Squares Mean (Standard Error); unit: kPCD/minutes
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
Number analyzed (Participants) | 9 | 6 | 8
kPCD/minutes | 267.12 (708.056) | 283.09 (871.664) | 221.74 (738.728)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg vs Placebo; Test type: Superiority; p < 0.05, ANCOVA — Adjustment for multiple comparisons were made using Dunnett's test at the overall alpha = 0.05 significance level; Fixed effects for treatment group (PCS12852 0.1 mg, PCS12852 0.5 mg, and Placebo) and type (IG or DG) and the baseline value as a continuous covariate

2. Primary Outcome: Change in Gastric Emptying Rate From Baseline Using t50 Metric for Gastric Emptying Rate
Description: Time for 50% gastric emptying (t50) metric assessed by the GEBT
Time Frame: ~28 days
Population: The change from baseline to Day 28 using the t50 metric was analyzed using an analysis of covariance (ANCOVA) model with fixed effects for treatment group and gastroparesis type (idiopathic gastroparesis [IG] or diabetic gastroparesis [DG]) and the baseline value as a continuous covariate. Only patients with a baseline and Day 28 value were included in the analysis. The parameters listed are the best comparison of the breath test as opposed to individual timepoints.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
Number analyzed (Participants) | 9 | 6 | 8
Minutes | -4.89 (12.320) | -26.64 (14.971) | -11.15 (12.365)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg vs Placebo; Test type: Superiority; p < 0.05, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Concentrations of PCS12852 in Plasma - Cmax
Description: PK parameters were estimated from concentration-time data using noncompartmental methods, as data permitted.
Time Frame: Day 1
Population: PK parameters were not calculated for patients with 2 or fewer detectable concentrations in their PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg
Number analyzed (Participants) | 7 | 7
ng/mL | 0.12211 (0.039216) | 0.59986 (0.329187)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg; Test type: Superiority; p < 0.05, Regression, Linear

4. Primary Outcome: Concentrations of PCS12852 in Plasma - AUC0-last
Description: PK parameters were estimated from concentration-time data using noncompartmental methods, as data permitted.
Time Frame: Day 1
Population: PK parameters were not calculated for patients with 2 or fewer detectable concentrations in their PK profile.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg
Number analyzed (Participants) | 7 | 7
h*ng/mL | 0.6331 (0.27524) | 3.0612 (1.58834)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg; Test type: Superiority; p < 0.05, Regression, Linear

5. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD
Description: Change from baseline in the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index Daily Diary (ANMS GCSI-DD). Scores range from 0-4 for the gastroparesis-related symptoms (nausea, early satiety, postprandial fullness, upper abdominal pain, and vomiting), with 4 meaning a worse outcome.
Time Frame: Day 7
Population: Scores were not able to be calculated for some patients in 0.5mg group due to 2 patients discontinuing.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
Number analyzed (Participants) | 8 | 6 | 8
score on a scale | -0.02 (0.141) | -0.69 (0.171) | -0.58 (0.138)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

6. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD
Description: Change from baseline in the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index Daily Diary. Scores range from 0-4 for the gastroparesis-related symptoms (nausea, early satiety, postprandial fullness, upper abdominal pain, and vomiting), with 4 meaning a worse outcome.
Time Frame: Day 14
Population: Scores were not able to be calculated for some patients in the 0.5mg group due to 2 patients discontinuing.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
Number analyzed (Participants) | 8 | 6 | 8
Units on a scale | -0.62 (0.218) | -1.06 (0.267) | -0.82 (0.210)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

7. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD
Description: as for outcome 6
Time Frame: Day 21
Population: Scores were not able to be calculated for some patients in the 0.5mg group due to 2 patients discontinuing.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
Number analyzed (Participants) | 8 | 6 | 8
Units on a scale | -0.57 (0.237) | -1.12 (0.290) | -0.91 (0.228)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

8. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD
Description: as for outcome 6
Time Frame: Day 28
Population: Scores were not able to be calculated for some patients in the 0.5mg group due to 2 patients discontinuing.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
Number analyzed (Participants) | 8 | 6 | 8
Units on a scale | -0.61 (0.254) | -1.48 (0.311) | -1.00 (0.244)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg vs Placebo; Test type: Superiority; p < 0.05, ANCOVA

9. Primary Outcome: Concentrations of PCS12852 in Plasma - AUC0-last
Description: PK parameters were estimated from concentration-time data using noncompartmental methods, as data permitted.
Time Frame: Day 28
Population: PK parameters were not calculated for patients with 2 or fewer detectable concentrations in their PK profile.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg
Number analyzed (Participants) | 7 | 5
h*ng/mL | 1.0987 (1.23183) | 7.4218 (7.10856)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg; Test type: Superiority; p < 0.05, Regression, Linear

10. Primary Outcome: Concentrations of PCS12852 in Plasma - Cmax
Description: PK parameters were estimated from concentration-time data using noncompartmental methods, as data permitted.
Time Frame: Day 28
Population: PK parameters were not calculated for patients with 2 or fewer detectable concentrations in their PK profile.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg
Number analyzed (Participants) | 7 | 5
ng/mL | 0.11984 (0.068770) | 0.48100 (0.255856)
Statistical Analysis 1: Comparison: PCS12852 0.1mg vs PCS12852 0.5mg; Test type: Superiority; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the Informed Consent Form was signed to the last study visit on Day 35.
Arm/Group | PCS12852 0.1mg | PCS12852 0.5mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 5/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCS12852 0.1mg (N=9) | PCS12852 0.5mg (N=8) | Placebo (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05270460/Prot_SAP_000.pdf